CLINICAL TRIAL: NCT02121769
Title: Protocol for Patients With Parenteral Nutrition Associated Liver Disease (PNALD) to Access Parenteral Fish Oil (Omegaven®) - Omegaven IND 122375
Brief Title: Omegaven Expanded Access Protocol
Status: No longer available | Type: Expanded Access
Sponsor: St. Luke's Health System, Boise, Idaho (Other)
Responsible Party: Principal Investigator, Tyler Burpee, MD, Principal Investigator, St. Luke's Health System, Boise, Idaho
Other Study IDs: Omegaven Expanded Access
Record Dates: First submitted 2014-04-21; First posted 2014-04-24 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Parenteral Nutrition Associated Liver Disease
Keywords: cholestasis; short bowel syndrome
MeSH Terms: conditions — Cholestasis; Short Bowel Syndrome | interventions — fish oil triglycerides

INTERVENTIONS:
Drug: Omegaven — 10% Omegaven 1g/kg/day, Intravenous by continuous infusion in conjunction with parenteral nutrition, until the patient no longer requires parenteral nutrition or until participation in the study is terminated.

SUMMARY:
Omegaven is an intravenous fat emulsion (IFE) comprised of omega-3 fatty acids derived from fish oil. It will be used in an open label compassionate use treatment protocol, as an alternative to soybean oil (omega-6), as the sole IFE source of parenteral nutrition in an effort to reduce and/or reverse parenteral nutrition associated liver disease. The study will evaluate the safety and efficacy of Omegaven use in pediatric patients with PN dependence and PNALD.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be PN dependent (unable to meet nutritional needs solely by enteral nutrition) and are expected to require PN for at least another 30 days
* Parenteral nutrition associated liver disease (PNALD) as defined as a direct bilirubin of ≥ 2 mg/dL on the last two consecutive bilirubins while on PN. Other causes of liver disease should be excluded. A liver biopsy is not necessary for treatment.
* Failed standard/conventional therapies to prevent progression of PNALD.
* Age newborn to 17 years of age
* Signed informed consent.

Exclusion Criteria:

* Allergy to eggs and/or shellfish
* Female who is pregnant or lactating
* Severe hemorrhagic disorder
* Other causes of chronic liver disease (Hepatitis C, Cystic fibrosis, biliary atresia, and alpha 1 anti-trypsin deficiency,)
* 18 years of age or older
* Parent/legally authorized representative is unwilling to consent.

Max Age: 17 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Burpee, MD, Principal Investigator — Pediatric Gastroenterology
Locations (1):
- St. Luke's Pediatric Gastroenterology, Boise, Idaho, United States